CLINICAL TRIAL: NCT06722547
Title: The Effects of Addition Respiratory Muscle Stretching Exercise for Improving Functional Exercise Capacity Fatigue and Quality of Life in Patients With Bronchiectasis Post-Tuberculosis Lung Disease
Brief Title: Respiratory Muscle Stretching Exercise for Improving Quality of Life of Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKFR-202411.04
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Bronchiectasis Post-Tuberculosis Lung Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Standard Pulmonary Rehabilitation) (Active Comparator): Aerobic exercise, PLB, ACBT, Education
  Interventions: Other: Standard PR
- Group B (Standard PR + RMS) (Experimental): Standard PR plus Respiratory Muscle Stretching
  Interventions: Other: Standard PR plus Respiratory Muscle Stretching

INTERVENTIONS:
Other: Standard PR — PLB, ACBT, Aerobic exercise, Education
  Arms: Group A (Standard Pulmonary Rehabilitation)
Other: Standard PR plus Respiratory Muscle Stretching — Standard PR plus Respiratory Muscle Stretching (RMS)
  Arms: Group B (Standard PR + RMS)

SUMMARY:
Bronchiectasis is a chronic condition often arising after the successful treatment of lung tuberculosis, leading to diminished functional exercise capacity, increased fatigue, and reduced quality of life. This randomized controlled trial aims to evaluate the efficacy of adding Respiratory Muscle Stretching (RMS) exercises to standard pulmonary rehabilitation in improving functional exercise capacity, reducing fatigue, and enhancing the quality of life in patients with bronchiectasis post-tuberculosis.

DETAILED DESCRIPTION:
Bronchiectasis, a long-term sequelae of lung tuberculosis, is characterized by permanent dilation and damage of the bronchi, resulting in reduced lung function, persistent fatigue, and significantly impaired quality of life. Standard pulmonary rehabilitation (PR) programs, which include aerobic exercises and breathing techniques like Pursed Lip Breathing (PLB) and the Active Cycle of Breathing Technique (ACBT), are known to offer symptomatic relief and functional improvements. However, the role of Respiratory Muscle Stretching (RMS) in this context has not been well explored.

This clinical trial will assess the impact of RMS, when combined with standard PR, on key outcomes including functional exercise capacity, fatigue, and overall quality of life in patients with bronchiectasis following tuberculosis treatment. The study will involve a parallel assignment of patients to either the standard PR group or the PR plus RMS group, with outcomes measured over a 6-week intervention period. The primary endpoints will include changes in 6-Minute Walk Test (6MWT) distances, Fatigue Severity Scale (FSS) scores, and Quality of Life (St. George's Respiratory Questionnaire) scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-59 years
* History of lung TB treatment
* Clinical or radiological diagnosis of bronchiectasis
* mMRC Dyspnea Scale grade 1-3

Exclusion Criteria:

* Pneumothorax Pleural effusion
* Neuromuscular disease
* Lung malignancy
* history of COVID-19

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity (6-Minute Walk Test) | 6 weeks
  The 6-Minute Walk Test (6MWT) is a simple, objective, and widely used assessment tool to evaluate an individual's functional exercise capacity. It measures the total distance a person can walk in six minutes on a flat, hard surface at their own pace, serving as an indicator of aerobic capacity and endurance. This test is particularly useful in patients with chronic respiratory or cardiovascular conditions as it reflects their ability to perform daily physical activities. Prior to the test, baseline measurements of blood pressure, heart rate, oxygen saturation, and dyspnea (using the Borg Dyspnea Scale) are recorded. During the test, participants are encouraged with standardized verbal prompts while allowed to rest if needed. The primary outcome is the total distance walked, with additional observations such as pauses, walking speed, and symptoms documented. The 6MWT easy to administer, and provides valuable insights into a patient's functional status, treatment efficacy, and prognosis

SECONDARY OUTCOMES:
Fatigue (Fatigue Severity Scale) | 6 weeks
  Fatigue, a common symptom in chronic conditions, is characterized by a subjective sense of physical and mental exhaustion that can interfere with daily functioning. The Fatigue Severity Scale (FSS) is a validated self-reported questionnaire designed to assess the impact of fatigue on a person's ability to perform routine activities. Comprising nine items, the FSS measures the severity of fatigue experienced over the past week, with responses ranging from 1 (strong disagreement) to 7 (strong agreement). A higher mean score indicates greater fatigue severity. The FSS is widely used in clinical and research settings for its reliability and ability to distinguish fatigue levels in patients with various conditions, including respiratory diseases, neurological disorders, and autoimmune diseases. It provides valuable insights into the extent of fatigue, helping guide interventions and monitor treatment outcomes.
Quality of Life (St. George's Respiratory Questionnaire) | 6 weeks
  The St. George's Respiratory Questionnaire (SGRQ) is a validated self-administered tool designed to assess health-related quality of life in patients with respiratory diseases. It consists of 50 items divided into three domains: Symptoms (frequency and severity of respiratory symptoms), Activity (activities limited by breathlessness), and Impacts (effects of the disease on daily life, including emotional aspects). Each domain and the total score range from 0 to 100, with higher scores indicating poorer health-related quality of life. The SGRQ provides a comprehensive evaluation of a patient's perception of their respiratory health, making it a valuable instrument for clinical trials, disease monitoring, and evaluating treatment outcomes. It has been translated into various languages, including Indonesian, ensuring reliability and validity across diverse populations.

CONTACTS AND LOCATIONS:
Overall Officials: Dian Marta Sari, MD., M.Sc., Ph.D, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Dr. M. Goenawan Partowidigdo Lung Hospital, Bogor, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allwood BW, Byrne A, Meghji J, Rachow A, van der Zalm MM, Schoch OD. Post-Tuberculosis Lung Disease: Clinical Review of an Under-Recognised Global Challenge. Respiration. 2021;100(8):751-763. doi: 10.1159/000512531. Epub 2021 Jan 5. PMID 33401266
- [Background] O'Leary CJ, Wilson CB, Hansell DM, Cole PJ, Wilson R, Jones PW. Relationship between psychological well-being and lung health status in patients with bronchiectasis. Respir Med. 2002 Sep;96(9):686-92. doi: 10.1053/rmed.2002.1330. PMID 12243314
- [Background] Sami R, Zohal M, Mohammadi N. Clinical Determinants of the Six-Minute Walk Test (6MWT) in Stable Non-Cystic Fibrosis Bronchiectasis Patients. Tanaffos. 2020 Dec;19(4):385-391. PMID 33959177
- [Background] Khosa C, Bhatt N, Massango I, Azam K, Saathoff E, Bakuli A, Riess F, Ivanova O, Hoelscher M, Rachow A. Development of chronic lung impairment in Mozambican TB patients and associated risks. BMC Pulm Med. 2020 May 7;20(1):127. doi: 10.1186/s12890-020-1167-1. PMID 32381002